CLINICAL TRIAL: NCT07021469
Title: Sound Origins: Assessment of the Acceptability and Accessibility of a Co-designed Music Therapy Intervention
Brief Title: Sound Origins Acceptability Study
Acronym: Soundorigins
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 355379
Record Dates: First submitted 2025-05-28; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Accessibility and Acceptability of Intervention
Keywords: music therapy; acceptablity; neonatal; NICU; palliative care; experienced based co-design

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent and staff participants (Experimental): Parents with infants with uncertain futures on admission to the neonatal unit and the nurses caring for them.
  Interventions: Other: Sound origins

INTERVENTIONS:
Other: Sound origins — Parents:
  1. Playlists created by parents with lived experience for parents to use as ideas for music they could use for themselves or with baby on the unit.
  2. Parent Journal: This journal provides a guide for using music and self-reflection. It also has the link for the playlists.
  3. 'Musical gifts' created with the support of a music therapist from external family/ friends to the baby on the unit.
  Nursing staff caring for families participating in the study:
  1. Nurses shared playlist. Suggested creation of 3 playlists for nursing staff to create their own shared playlist using their music.
  2. 'Ask me' badges. These badges are optional for nurses to wear during their shifts but will act as a symbol to parents that their nurse is available to speak to about music.
  Other Names: Sound origins music therapy approach; Neonatal music therapy intervention

SUMMARY:
The goal of this study is to assess the acceptability and accessibility of a co-designed music therapy intervention for parents with infants with uncertain futures and nursing staff on the neonatal unit. The main questions it aims to answer are:

1. To assess the acceptability and accessibility of the co-designed music therapy intervention
2. To assess the frequency of recruitment and retention of the participants
3. To assess the feasibility of the creation and sharing of a musical gift within 1 week
4. To assess the appropriateness of the timeframe for interview of parents who experience neonatal death during the study timeframe.

Participants will test an intervention comprising of:

1. Playlists created by parents with lived experience for parents to use as ideas for music they could use for themselves or with baby on the unit. This is shared via QR code in a journal and on the study website which will be provided at the time of the consent.
2. Parent Journal: This journal provides a guide for using music and self-reflection. It also has the link for the playlists.
3. 'Musical gifts' created with the support of a music therapist from external family/ friends to the baby on the unit. Contact will be on MsTeams with individual age 18 or over or supported by an adult. Music will be created by contact to send direct to family on the neonatal unit as a voice note. If requested the family may send a voice note to the music therapist to then add to to make more complex music using 'Audacity' software to then be returned to the contact via 'we transfer' for approval before sharing with the family on the unit.
4. Nurses shared playlist: This is a playlist for nursing staff to create their own shared playlist using their music.
5. 'Ask me' badges. These badges are optional for nurses to wear during their shifts but will act as a symbol to parents that their nurse is available to speak to about music

DETAILED DESCRIPTION:
Testing a co-designed music therapy intervention:

This study will aim to test a co-designed music therapy interventions with 12 parents of 12 infants with uncertain futures at University College London hospital and the nurses that care for them during this period.

Parents will be approached by the lead researcher, research nurse or lead consultant about participating in the study. They will be given information sheets outlining what will be expected and the potential burdens and benefits of taking part. They will be given 24hrs to consider the study before providing consent. The lead researcher will then approach to gain consent and answer any questions on the study. If consent is given, the cot side nurse will provide the family with the journal and make a referral to music therapy. A meeting with the unit music therapist will then be made and the following discussed:

1. contact with a nominated person off the unit to create a musical gift for the baby (external contact will need to be age 18 or over, siblings/ children can be included if supported by an adult). Meeting held via MSTeams.
2. explanation of a website and parent playlists
3. a journal

After the music therapist has worked with the external contact and a musical gift created (likely to be a lullaby) it will be sent to the family either by the family contact or the music therapists as preferred by the parent. On day 7 of the study the music therapist will check in with the parent on the unit to review the materials and offer further support. Journal entries will not be shared with any member of staff or the researcher unless parents wish to. Parents can then chose to continue support or use the resources independently.

During the study period parents will be asked to complete questionnaires assessing psychological safety (Neuroception of psychological safety scale NPSS-G). These will be completed on the unit on day 1 and 16 of the study via hardcopy. Once completed, parents can leave with the reception in a sealed envelope (provided). This will then be stored in a locked research cabinet until the lead research is able to collect. Separately, nursing staff involved in the care of these babies will be encouraged to build a shared playlist to support staff relationships and regulation through music. They will be sent a digital link to the website which gives instruction and guide to engagement with families through music as well as advise on building a staff playlist. They will also be provided with 'ask me' badges to wear to signal their availability to parents that they are happy to engage in conversation about the parents use of music and the value of certain music to their family.

Evaluation of acceptability:

At the end of the study period (3 weeks) parents will be asked to complete an acceptability survey and attend a short interview. Where a baby has died parents will be contacted 6 weeks after the death to consent their continued participation in the study and completion of the survey and interview. The lead researcher will contact parents to arrange a time for a short interview either at the parents home or at a University College London Hospital research room to discuss the acceptability of the intervention further. Similarly health care professionals will also be ask to complete an acceptability survey at the end of the intervention being testing on the unit (4 months) and encouraged to give feedback on their use of the playlist and the 'ask me' badges. Prior to completing the questionnaire they will be required to complete a consent form where they can tick if they would like to be contacted to participate in an online focus group to discuss their experiences further. Those who chose to do this will be provided with an overview of the topics for discussion prior to the group.

Celebration event:

A celebration event will be held at King's Place, London to celebrate the development of the intervention and the value of the engagement from everyone who has been involved at all stages. Everyone involved at any stage of the research will be invited to this event. It will also be extended to healthcare professionals and family support charities.

ELIGIBILITY:
Inclusion Criteria:

Parent inclusion criteria:

1. 18+ years
2. Has an infant diagnosed with a condition meeting the infant inclusion criteria on admission to the unit (see below)
3. Can give informed consent

Healthcare professional inclusion criteria:

1. Nursing professional working with or providing support to parents with infants diagnosed with a life limiting condition involved in the study
2. Part time, full time on UCLH neonatal unit
3. Any grade

Infant inclusion

In accordance with Together for short lives neonatal palliative care guidelines any parent who has an infant meeting the following criteria whilst on the neonatal unit will be eligible for the intervention:

Category 1: Life-threatening conditions for which curative treatment may be feasible but can fail Provision of palliative care services may be necessary when treatment fails or during an acute crisis, irrespective of the duration of threat to life. On reaching long-term remission or following successful curative treatment there is no longer a need for palliative care services. Examples: extreme prematurity, severe necrotising enterocolitis, congenital heart disease.

Category 2 Conditions where premature death is inevitable. There may be long periods of intensive treatment aimed at prolonging life and allowing participation in normal activities. Example: chromosomal abnormality, severe spina bifida, bilateral multi-cystic dysplastic kidneys, bilateral renal agenesis.

Category 3 Progressive conditions without curative treatment options Treatment is exclusively palliative and may commonly extend over many years. Example: skeletal dysplasia, severe neuromuscular disorders.

Category 4 Irreversible but non-progressive conditions causing severe disability, leading to susceptibility to health complications and likelihood of premature death. Example: severe hypoxic ischaemic encephalopathy.

Exclusion Criteria:

Parent exclusion criteria

1. <18+ years
2. Acute mental health diagnosis e.g schizophrenia, psychosis
3. Substance abuse
4. Does not have an infant meeting inclusion criteria
5. Unable to provide consent

Healthcare professional exclusion criteria

1. not working with or providing support to parents with infants diagnosed with a life limiting condition
2. agency staff

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability Questionnaire | Parents will be assessed after completing the intervention for 3 weeks. Staff will complete the questionnaire at the end of the full study duration. This will be either after 4 months or when 12 parents have participated whichever is first.
  A non-validated questionnaire developed by the researchers will assess the acceptability of the intervention based on domains from Sekon's Theoretical Framework of Acceptability. The framework includes the following domains: Affective attitude, burden, ethicality, perceived effectiveness, opportunity cost, intervention coherence, self-efficacy. These will be assessed through one questionnaire.

SECONDARY OUTCOMES:
Neuroception of psychological safety scale- NPSS | Days 1 and 16
  Assessment of parent perceived psychological safety: Participants rate how well statements describe their feelings on a likert scale (strongly disagree =1 up to Strongly Agree=5). Higher scores relate to higher levels of perceived psychological safety.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Robert, PhD, Study Chair — King's College London; Kirsty Jane, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - Kings College London, London, Professor
  - University College London Hospital Neonatal Unit, London

IPD SHARING:
Plan to Share IPD: No
This is a small scale acceptability testing study as part of the lead researchers PhD.

REFERENCES:
- [Background] Jane K, Wood D, Gallagher K, Livermore P, Shoemark H, Robert G. Parents' experiences of psychotherapeutic support on the neonatal unit: A mixed methods systematic review to inform intervention development for a multicultural population. Nurs Crit Care. 2025 May;30(3):e13194. doi: 10.1111/nicc.13194. Epub 2024 Oct 28. PMID 39467007
- [Background] Standley J. Music therapy with premature infant: Research and developmental interventions. Music Therapy Perspectives. 2003;23(1):76-8.
- [Background] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Background] Flaks MK, Malta SM, Almeida PP, Bueno OF, Pupo MC, Andreoli SB, Mello MF, Lacerda AL, Mari JJ, Bressan RA. Attentional and executive functions are differentially affected by post-traumatic stress disorder and trauma. J Psychiatr Res. 2014 Jan;48(1):32-9. doi: 10.1016/j.jpsychires.2013.10.009. Epub 2013 Oct 22. PMID 24199652
- [Background] Al Maghaireh DF, Abdullah KL, Chan CM, Piaw CY, Al Kawafha MM. Systematic review of qualitative studies exploring parental experiences in the Neonatal Intensive Care Unit. J Clin Nurs. 2016 Oct;25(19-20):2745-56. doi: 10.1111/jocn.13259. Epub 2016 Jun 3. PMID 27256250
- [Background] Fraser. L. G-SD, Jarvis. D., Norman. P., Parslow. R., . 'Make Every Child Count' Estimating current and future prevalence of children and young people with life-limiting conditions in the United Kingdom. Together for Short Lives. 2020.
- [Background] NCMD. NCMD Second Annual Report. Child Death Review Data. 2021.
- [Background] Dickson G. A Perinatal Pathway for Babies with Palliative Care Needs, 2nd Edition. Together for Short Lives. 2019.
- See also: Sound Origins Study, King's College London — https://www.kcl.ac.uk/research/sound-origins-connecting-through-voice